CLINICAL TRIAL: NCT01558934
Title: A Pilot, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Electrocardiographic Effects of Lofexidine When Administered Orally to Methadone Maintained Adult Subjects
Brief Title: Pilot Study of Lofexidine and Methadone Pharmacodynamic Interaction in Methadone Maintained Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-LX1-1005-1; 1U01DA030916-01 (NIH)
Record Dates: First submitted 2012-02-14; First posted 2012-03-20 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Opioid Dependence; Methadone Withdrawal Syndrome
Keywords: lofexidine; methadone; interaction; pharmacodynamic; ECG; QTc
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lofexidine Titration in Methadone Maintained Subjects (Experimental): Methadone maintained subjects will be titrated on lofexidine up to the target therapeutic dose of 0.8 mg QID or to the highest level tolerated. Following this initial titration attempt, all subjects will have their methadone dose reduced by 50% and lofexidine titration efforts will resume. If the therapeutic dose is not reached under 50% methadone reduction conditions, the methadone dose will be further reduced to 0 mg for 2 days followed by reintroduction of 25% of the starting dose on the 3rd day, and on such 3rd day lofexidine titration will resume again.
  Interventions: Drug: Lofexidine HCl

INTERVENTIONS:
Drug: Lofexidine HCl — Lofexidine HCl 0.2 mg tablets titrated in ascending doses of 0.2 mg QID (e.g. Day 1 0.2 mg QID, Day 2 0.4 QID, etc)as described in the treatment arm.

SUMMARY:
The primary objective of this study is to assess QTc (an interval of the heart rhythm) interaction effects between lofexidine and methadone. The secondary objectives of the study are to evaluate the safety and tolerability of lofexidine by evaluating and monitoring pharmacokinetics (amounts of drug in the blood), vital signs (heart rate and blood pressure) and adverse events (side effects) when co-administered with methadone; and to describe effects on opiate withdrawal when lofexidine is introduced following a 50% or 100% methadone dose reduction, as required to elicit a withdrawal response. The investigators hypothesize that while both agents are known to prolong the QTc interval, the combination of the drugs will not create an additive effect which creates a significant safety concern. The investigators further hypothesize that subjects will be able to tolerate the therapeutic dose of lofexidine (0.8 mg four times daily) when the methadone maintenance dose is lowered to elicit withdrawal.

DETAILED DESCRIPTION:
This will be an open-label multiple ascending dose study to assess the safety, tolerability, and electrocardiographic effects of lofexidine in 6 methadone-maintained adult subjects. The study will include a Screening Visit, an Inpatient Treatment Visit, and a Follow-Up Visit.

Subjects who are on a stable dose of methadone (80 - 120 mg/day) and who satisfy inclusion and exclusion criteria will be eligible for the study. Within 21 days of the Screening Visit, subjects will report to the inpatient study facility to begin the Inpatient Treatment Visit which will last between 10 to 27 days. This visit will include an inpatient check-in (1 day), Methadone Baseline (1 day), Initial Lofexidine Titration (up to 4 days), 1, 2 or 3 Lofexidine Plateaus (2 days each), Methadone Reduction (up to 11 days), and Methadone Re-Titration and Discharge (up to 4 days). The order of steps subjects will proceed through during the Inpatient Treatment Visit will vary depending on subjects' ability to titrate to a 0.8 mg QID dose of lofexidine and whether or not they experience opiate withdrawal during methadone reduction. Diagrams for the three scenarios that can occur with lofexidine titration are located in Figure 1, 2, and 3 in the body of the protocol.

During the Methadone Baseline phase subjects will take a single daily dose of methadone at 1 PM and undergo baseline study assessments including electrocardiogram (ECG) monitoring and blood collection for methadone pharmacokinetics. The next day subjects will proceed to the Initial Lofexidine Titration phase. Subjects will continue using their baseline methadone dose. Lofexidine will be initiated at 0.2 mg QID and titrated in daily increments of 0.2 mg QID to a total dose of 0.8 mg QID (3.2 mg/day), if tolerated by the subject. Lofexidine doses will escalate daily unless at any point the subject meets protocol-defined dose hold criteria (described below), which will trigger a reduction in dose to the previous highest tolerated dose. Once subjects have titrated to the 0.8 mg QID dose or once the highest tolerated dose of lofexidine has been determined, they will proceed to a 2-day Lofexidine Plateau phase during which they will continue to receive their methadone maintenance dose. If the subject is not able to titrate up to 0.8 mg QID, the subject will continue to receive their highest tolerated dose in equal increments (eg, 0.2, 0.4, or 0.6 mg QID at 8AM, 1PM, 6PM, 11PM) for both days of the plateau. If the subject tolerates 0.8 mg QID lofexidine, on the first day they will receive 0.8 mg QID lofexidine according to the normal dosing schedule. On the second day the lofexidine dosing schedule will be modified with subjects receiving a 0.2 mg increase of the 1 PM lofexidine dose (1 mg dose) and a 0.2 mg reduction in the subsequent lofexidine dose (0.6 mg dose) with the other 2 doses of 0.8 mg (total dose of 3.2 mg/day). On the second day of the Lofexidine Plateau phase, subjects will undergo electrocardiogram (ECG) monitoring and blood collection for methadone and lofexidine pharmacokinetics.

Subjects who are unable to titrate to the 0.8 mg QID lofexidine dose while receiving their full dose of methadone will undergo a methadone dose reduction of 50%, or if necessary a dose reduction of 100%, and will continue lofexidine titration by adding an incremental 0.2 mg QID to the previously established tolerated dose up to the maximum 0.8 mg QID dose. During these subsequent titration attempts lofexidine doses will escalate daily unless in any event a subject meets protocol defined dose-hold criteria (described below), which will trigger a reduction in dose to the previous highest tolerated dose and will require the Lofexidine Plateau procedures described above to be repeated while maintaining the subject on their newly reduced methadone dose (eg, 50% of their maintenance dose and, if 0.8 mg QID is not achieved at the first reduction, again at 0% of their maintenance dose for 2 days followed by reinstatement of 25% of their starting dose).

Subjects who are able to titrate to the 0.8 mg QID lofexidine dose while receiving their full dose of methadone will continue to receive the maximum lofexidine dose while undergoing a 4 day Methadone Reduction at 50% of their maintenance dose to evaluate lofexidine's impact on the withdrawal syndrome.

During Methadone Reduction (whether for subjects entering an experimental 4-day 50% withdrawal phase at the tolerated 0.8 mg QID lofexidine dose or for subjects continuing lofexidine titration at 50% and 100% methadone reductions), assessments of opiate withdrawal will be performed using the Clinical Opiate Withdrawal Scale (COWS) and the Short Opiate Withdrawal Scale (SOWS).

Following completion of the Lofexidine Plateau (repeated as necessary) and Methadone Reduction, subjects will begin the Methadone Re-Titration and Discharge phase during which lofexidine will be discontinued (except to treat withdrawal symptoms as necessary) and methadone will be re-titrated to the starting dose (or to a higher or lower dose relative to baseline as medically indicated at the discretion of the investigator). Following successful methadone titration and completion of study assessments, subjects will be discharged from the inpatient study clinic.

Subjects will return to the study clinic for a follow-up visit 7 days (±2 days) following clinic discharge for safety follow-up and adverse event collection. Subjects will be discharged from the study at this time unless they are medically unstable on their dose of methadone. Subject may be medically followed at a regular interval, as determined by the investigator, until the subject is considered sufficiently stable for study discharge.

Subjects who withdraw consent or meet any one of the following study termination criteria prior to completion of the study will be withdrawn:

1. Cardiovascular events including the following:

   1. Systolic blood pressure <70 mmHg and >20% below screen value;
   2. Diastolic blood pressure <40 mmHg and >20% below screen value:
   3. Heart rate <40 bpm and >20% below screen value;
   4. QTc >500 msec or >25% above screen value for both males and females;
   5. Syncope. *ECGs and vital signs may be repeated as appropriate to confirm values and rule out extraneous results.
2. Serious medical problems thought to be related or unrelated to the study medications.
3. Intercurrent illness or medical complications that, in the opinion of the site investigator, preclude safe administration of study medications.

At the time of termination from the study, subjects will be discontinued from lofexidine; however, they may remain inpatient for up to 4 days while their methadone maintenance dose is re-titrated to their pre-study maintenance dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and/or female, 18 to 60 years of age (inclusive)
2. Receiving methadone maintenance treatment for opioid dependence at a stable once-daily dose of 80-120 mg for at least 4 weeks prior to check-in for the Inpatient Treatment Visit.
3. Body mass index ≥ 18 and ≤ 35 (kg/m2).
4. Normal screening results or abnormal results that have been deemed by the Investigator as clinically insignificant.
5. Able to understand and willing to sign an informed consent form (ICF).
6. Females practicing adequate birth control or non-childbearing potential. Medically acceptable birth control methods for this study include intrauterine device (IUD); vasectomized partner (minimum of 6 months); post-menopausal (at least 2 years); surgically sterile (at least 6 months); double barrier (diaphragm with spermicide, condoms with vaginal spermicide); abstinence; implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months prior to study dosing and throughout the study duration; and oral, patch and injected hormonal contraceptives or vaginal hormonal device (ie, NuvaRing®) in use for at least 3 consecutive months prior to study dosing and throughout the study duration.

Exclusion Criteria:

1. Abnormal cardiovascular exam at screening and before randomization, including any of the following:

   * clinically significant abnormal electrocardiogram (ECG) (eg, significant first degree atrioventricular block, second or third degree heart block, clinically significant arrhythmia, or QTc interval (machine read) greater than 450 msec for males and greater than 470 msec for females)* heart rate < 55 bpm or symptomatic bradycardia*
   * systolic blood pressure (SBP) < 95 mmHg or symptomatic hypotension*
   * diastolic blood pressure (DBP) < 65 mmHg*
   * blood pressure (BP) > 155/95 mmHg*
   * change in orthostatic SBP, DBP, or heart rate >25% below recumbent values
   * prior history of myocardial infarction (MI) or evidence of prior MI on ECG* *ECGs and vitals may be repeated as appropriate in order to confirm values and rule out extraneous results.
2. History or presence of significant cardiovascular, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, psychiatric, neurologic, or dermatologic disease.
3. History or presence of any degree of chronic obstructive pulmonary disease.
4. History of suicidal ideations or depression requiring professional intervention including counseling or antidepressant medication.
5. Positive drug (urine)/alcohol (breath) test at Screening Visit or check-in to the Inpatient Clinic Visit excluding methadone. Subjects who have a positive test for heroin and benzodiazepines at the Screening Visit may be enrolled if the test is negative at check-in to the Inpatient Treatment Visit. Subjects who have a positive test for heroin or benzodiazepines at the Screening Visit must sign an ICF at check-in to the Inpatient Clinic Visit.
6. Receiving methadone for pain management.
7. Positive test for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg). Subjects with a positive test for hepatitis C antibodies (HCV) may be enrolled if subject is asymptomatic.
8. Estimated creatinine clearance < 80 mL/minute at screening (Cockcroft-Gault formula).
9. AST, ALT, or alkaline phosphatase > 3.0 x upper limit of normal at screening or check-in.
10. Amylase or lipase > 1.5 x upper limit normal at screening or check-in.
11. History of hypotension.
12. History of hypersensitivity or allergy to clonidine or any clonidine analogue.
13. Use of any new prescription medication within 12 days prior to check-in.
14. Use of any over-the-counter medication, including herbal products, within the 5 days prior to check-in. Up to 2 grams per day of acetaminophen is allowed at the discretion of the PI/PI"s designee.
15. Use of any drug known to affect QTc within 30 days prior to check-in (tobacco excluded).
16. Blood donation or significant blood loss within 30 days prior to check-in.
17. Plasma donation within 7 days prior to check-in.
18. Participation in another clinical trial within 30 days prior to check-in.
19. Females who are pregnant or lactating.
20. Any other condition or prior therapy, which, in the opinion of the Investigator, would make the subject unsuitable for this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes in QTc Interval | baseline and at each escalating lofexidine dosing plateau day 3 (participant time in the study will vary based on tolerability but each dose plateau will be evaluated after 3 days at any given dose level)
  The ECG analysis will be conducted by a central laboratory under blinded review. QTc intervals at baseline (methadone maintenance dose only) will be compared to a time matched profile at each increasing lofexidine dose (as tolerated by the subjects), both before and after a withdrawal response is elicited.

SECONDARY OUTCOMES:
Change from Baseline in the Short Opioid Withdrawal Scale (SOWS) | baseline and daily assessments during methadone withdrawal phases (participant time in withdrawal will vary based on lofexidine tolerability, however on average subjects will be in a methadone withdrawal phase of the study for approximately 10 days)
  SOWS Scores at Baseline (representing when a patient is on his/her normal methadone maintenance dose when withdrawal should be minimal or zero) will be compared to SOWS Scores during methadone reduction phases of the study to determine how the intervention is affecting withdrawal. Smaller changes from baseline indicate better control of withdrawal symptoms.
Change from Baseline in the Clinical Opiate Withdrawal Scale (COWS) | baseline and daily assessments during methadone withdrawal phases (participant time in withdrawal will vary based on lofexidine tolerability, however on average subjects will be in a methadone withdrawal phase of the study for approximately 10 days)
  COWS Scores at Baseline (representing when a patient is on his/her normal methadone maintenance dose when withdrawal should be minimal or zero) will be compared to COWS Scores during methadone reduction phases of the study to determine how the intervention is affecting withdrawal. Smaller changes from baseline indicate better control of withdrawal symptoms.
Methadone Area Under the Curve (AUC) | Baseline pre-dose, 2, 3, 4, 5, 6, 10 and 24 hours; plateau days pre-dose, 0.5, 1 , 2, 3, 4, and 5 hours post dose
  AUC will be calculated for methadone at baseline and at each escalating lofexidine dosing plateau day 3 (participant time in the study will vary based on tolerability but each dose plateau will be evaluated after 3 days at any given dose level)
Lofexidine Area Under the Curve (AUC) | plateau days pre-dose, 0.5, 1 , 2, 3, 4, and 5 hours post dose
  AUC will be calculated for lofexidine at each escalating lofexidine dosing plateau day 3 (participant time in the study will vary based on tolerability but each dose plateau will be evaluated after 3 days at any given dose level)
Change in Vital Signs | baseline and each day the lofexidine dose is escalated (participant time in the study will vary based on tolerability, however the participants will be exposed to up four different lofexidine doses (escalating from 0.2 QID to 0.8 mg QID)
  Vital signs of subjects on methadone alone (baseline) will be compared to participant vital signs while taking methadone and the range of studied lofexidine doses.
Change in Adverse Events | baseline and each day the lofexidine dose is escalated (participant time in the study will vary based on tolerability, however the participants will be exposed to up four different lofexidine doses (escalating from 0.2 QID to 0.8 mg QID)
  Adverse Events in subjects on methadone alone (baseline) will be compared to participant adverse events while taking methadone and the range of studied lofexidine doses.

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Gorodetzky, MD, PhD, Study Director — US WorldMeds; James A Longstreth, PhD, Study Director — US WorldMeds
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States